CLINICAL TRIAL: NCT03826953
Title: Allergy UK Research and Development Nurse. Developing and Evaluating the Impact of a Nurse-led Primary Care-based Allergy Clinic in NHS Lothian: a Mixed Methods Pilot Study
Brief Title: Allergy UK Research and Development Nurse Project
Acronym: ALLUKN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Allergy UK (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AC17008
Record Dates: First submitted 2017-05-22; First posted 2019-02-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2019-01

CONDITIONS: Allergy
Keywords: nurse led allergy clinic
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: The study is to determine the feasibility of a nurse led allergy clinic, delivered by specialist allergy nurse in primary care, using a hub and spoke model for the delivery of the clinic, the hub being the 'host' centre of GP practice and the spokes being the local / neighbouring GP practices that refer into the 'host' centre. Participants will be identified and recommended through their usual health care provider and referred into the clinic. Data will be collected through a mixed methods approach using questionnaires, interviews and national and locally held data to evaluate the effectiveness of the clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nurse led allergy clinic (Other): nurse led allergy clinic
  Interventions: Other: Nurse Led Allergy Clinic

INTERVENTIONS:
Other: Nurse Led Allergy Clinic — Project to investigate if it is feasible to establish a nurse-led primary care-based allergy clinic intervention in NHS Lothian, and to understand the acceptability and estimate the impact of this service on improving access and outcomes in patients with allergic conditions.WE will undertake a mixed-methods longitudinal evaluation of the community-based nurse-led allergy clinic.

SUMMARY:
The aim of the research project is to develop, deliver and assess the feasibility of a nurse-led allergy clinic in primary care, taking into account population, geographical area and needs of healthcare in the area chosen. It is widely acknowledged that the majority of cases of mild to moderate allergy could be adequately dealt with in primary care, by a healthcare professional with the appropriate expertise and knowledge of allergy. The provision of allergy care in the community could potentially have a beneficial impact on health care and patient outcomes.

The project will comprise the set up and delivery of a nurse led allergy clinic in primary care and use a mix of qualitative and quantitative methods to evaluate the feasibility of the clinic. This will include the use of a series of validated questionnaires e.g. satisfaction, condition specific quality of life and economic cost questionnaires, as well as face to face interviews.

The research will collect data to see if this clinical intervention is feasible and allow audit of the clinical intervention. This will also enable the researchers to understand patients lived experiences of accessing allergy care and the effect of allergy on quality of life and impact of allergy care.

DETAILED DESCRIPTION:
The study will consist of the development and delivery of a nurse led clinical intervention to provide allergy care in the community within the NHS Lothian primary care setting. The clinical intervention will see the allergy nurse provide clinical care to patients with a specified range of allergic conditions and provide diagnosis and immediate management where appropriate.

The clinical component of the research project will consist of a pilot nurse led allergy clinic, provided by one specialist nurse twice a week across two different GP surgeries within NHS Lothian, GPs from across 12 practices will be encouraged to refer into the pilot allergy clinic.

The referring health care professional will advise participants and their carers that the nurse led allergy clinic has been set up as part of a research project and participants will be asked if they wish to consent to take part in the research study. Feedback on the pilot clinic will be gathered to find out if the pilot clinic is acceptable to participants (satisfaction questionnaire), to find out if the clinic has made any improvement to quality of life (condition specific quality of life questionnaire) and if there is any cost impact (cost questionnaire).

Participants The initial consultation - explanation of research project and written informed consent obtained.

The nurse practitioner will:

* Take a thorough allergy clinical history including examination of the participant as necessary and identify what clinical care is required,
* Carry out any investigations that are required eg Skin prick testing to common food and aeroallergens.
* Give advice both written and verbal to support the management of allergies, including demonstration of medical devices e.g. adrenaline auto injectors, inhalers etc.
* Prescribe any necessary medication
* Provide a written summary of the consultation and any prescribed medication.

Participants will complete a series of three questionnaires, satisfaction, condition specific quality of life and cost questionnaires.

Follow up appointments where deemed appropriate will be conducted by telephone using a specified protocol. Where this is not appropriate face to face reviews will be arranged during clinic time. While short term follow-ups will be provided, there are no facilities to offer long term follow up for participants attending the allergy clinic under this pilot and all participants will return to their health care professional for follow up and long term management. If the participant has complex allergies or requires specialist intervention the participant will be advised that they will require referral into secondary care.

As part of the research project an email support service will be set up to support the health care professionals involved in the project.

The study will utilize a combination of qualitative and quantitative methods to evaluate the clinical intervention at baseline and at six weeks to determine the feasibility of the clinic and patient outcomes with this clinical intervention.

The tools available to the researcher include a series of validated surveys including patient and clinician satisfaction surveys, condition specific quality of life and economic cost to patient.

Interviews In addition face to face interviews will be offered to a subset of participants to enable further understanding of their perspective and experiences of the nurse-led allergy clinic. This will be to see if this intervention is feasible and improves patient care.

The views of health care professionals and practice managers referring into this clinic will also be sought using a satisfaction questionnaire and qualitative interviews at 12 weeks after the start of the clinic and 10-12 months from the end of the project.

Data on allergy will be requested from GP practices and NHS Information services Division (ISD) for quantitative analysis at baseline and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

All children, young people and adults who fit the selection criteria from across all the practices can be referred to the allergy clinic.

All patients and parents / carers where appropriate must be deemed capable of giving informed consent to take part in the research project.

* Infants under two with suspected food allergy
* Infants under two with moderate-to-severe eczema not responding to standard treatment.
* Children and young people (up to 16 years of age) with suspected allergic rhinitis symptoms that are unresponsive to a combination of oral antihistamines and nasal steroids
* Young people and adults (from 16 years of age) with a history of anaphylaxis or suspected anaphylaxis

Exclusion Criteria:

* Over 2 years of age with delayed type food allergy presenting primarily with gastrointestinal symptoms
* Over 2 years of age with confirmed non IgE-mediated symptoms including food intolerances, coeliac disease etc.
* Single urticarial reactions without an obvious triggers
* Non-allergic chronic urticaria
* Drug allergy
* Well controlled allergic rhinitis, asthma or atopic eczema
* Mild-to-moderate atopic eczema without an obvious allergic trigger
* Localised insect sting reactions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
To find out if a nurse-led clinic in primary care is feasible measured using a validated satisfaction questionnaire,in patients | 3 year feasibility study
  The questionnaire will measure the number of patients who had a positive or negative experience within the clinic using the satisfaction questionnaire at initial consultation then again at review
To find out if a nurse-led clinic in primary care is feasible measured using a validated satisfaction questionnaire in primary care | 3 year feasibility study
  The questionnaire will measure health care professionals experience of referring patients into the clinic using the satisfaction questionnaire
To find out if a nurse-led clinic in primary care is feasible measured using a validated health economics survey | 3 year feasibility study
  The Health economics survey will measure the cost of attending the clinic in terms of travel and loss of working or education hours required to attend the clinic.
To find out if a nurse-led clinic in primary care is feasible measured using qualitative interviews | 3 year feasibility study
  Qualitative interviews will be used to find out patients and health care professionals experience of using the nurse led allergy clinic, interview will be transcribed and analysed using Nvivo.

SECONDARY OUTCOMES:
Measure quality of life in patients using validated disease specific quality of life questionnaires Infants Dermatology Quality of Life Index IDQOL | 3 Years
  Will be used to determine if there is an improvement in a patients quality of life after attending the clinic this will be assessed using a validated quality of life questionnaire specifically designed for infants with dermatology. Scoring system is via a 4 point satisfaction scale none (no impact) =0 severe = 4
Measure quality of life in patients validated disease specific quality of life questionnaires Mini Rhinitis Quality of Life Questionnaire (mini RQLQ) | 3 Years
  Will be used to determine if there is an improvement in a patients quality of life after attending the clinic this will be assessed using a validated quality of life questionnaire to measure the impact of allergic rhinitis using a satisfaction scoring system no impact 0 - extreme = 4
Measure quality of life in patients validated disease specific quality of life questionnaires Food Allergy Quality of Life Questionnaire - Adult Form - (FAQLQ - AF) | 3 Years
  Will be used to determine if there is an improvement in a patients quality of life after attending the clinic this will be assessed using a validated quality of life questionnaire specifically designed for adults with food allergy, using a specially designed nummular 6 point rating scoring system where 0== no impact 3= moderate impact and 6 = extreme impact on quality of life
Measure quality of life in patients validated disease specific quality of life questionnaires Food Allergy Quality of Life Questionnaire - Teenagers Form (FAQLQ - TF) | 3 Years
  Will be used to determine if there is an improvement in a patients quality of life after attending the clinic this will be assessed using a validated quality of life questionnaire specifically designed for teenagers with food allergy. Scoring system using a specially designed nummular 6 point rating scoring system where 0== no impact 3= moderate impact and 6 = extreme impact on quality of life
Measure quality of life in patients validated disease specific quality of life questionnaires Food Allergy Quality Of Life Questionnaire - Parents Form (FAQLQ - PF) | 3 Years
  Will be used to determine if there is an improvement in a patients quality of life after attending the clinic this will be assessed using a validated quality of life questionnaire specifically designed for parents with children under 12 with food allergy. Scoring system using a specially designed nummular 6 point scoring system where 0== no impact 3= moderate impact and 6 = extreme impact on quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Sheikh, Principal Investigator — University of Edinburgh
Locations (1):
- University Of Edinburgh Health Centre, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anandan C, Gupta R, Simpson CR, Fischbacher C, Sheikh A. Epidemiology and disease burden from allergic disease in Scotland: analyses of national databases. J R Soc Med. 2009 Oct;102(10):431-42. doi: 10.1258/jrsm.2009.090027. PMID 19797601
- [Background] Ben-Shoshan M, Soller L, Harrington DW, Knoll M, La Vieille S, Fragapane J, Joseph L, St Pierre Y, Wilson K, Elliott SJ, Clarke AE. Eczema in early childhood, sociodemographic factors and lifestyle habits are associated with food allergy: a nested case-control study. Int Arch Allergy Immunol. 2015;166(3):199-207. doi: 10.1159/000381829. Epub 2015 Apr 22. PMID 25926095
- [Background] Cummings AJ, Knibb RC, King RM, Lucas JS. The psychosocial impact of food allergy and food hypersensitivity in children, adolescents and their families: a review. Allergy. 2010 Aug;65(8):933-45. doi: 10.1111/j.1398-9995.2010.02342.x. Epub 2010 Feb 22. PMID 20180792
- [Background] Dhami S, Sheikh A. Estimating the prevalence of aero-allergy and/or food allergy in infants, children and young people with moderate-to-severe atopic eczema/dermatitis in primary care: multi-centre, cross-sectional study. J R Soc Med. 2015 Jun;108(6):229-36. doi: 10.1177/0141076814562982. Epub 2015 Jan 7. PMID 25567768
- [Background] Gupta R, Sheikh A, Strachan DP, Anderson HR. Burden of allergic disease in the UK: secondary analyses of national databases. Clin Exp Allergy. 2004 Apr;34(4):520-6. doi: 10.1111/j.1365-2222.2004.1935.x. PMID 15080802
- [Background] Jutel M, Angier L, Palkonen S, Ryan D, Sheikh A, Smith H, Valovirta E, Yusuf O, van Wijk RG, Agache I. Improving allergy management in the primary care network--a holistic approach. Allergy. 2013 Nov;68(11):1362-9. doi: 10.1111/all.12258. Epub 2013 Oct 11. PMID 24117436
- [Background] Levy ML, Walker S, Woods A, Sheikh A. Service evaluation of a UK primary care-based allergy clinic: quality improvement report. Prim Care Respir J. 2009 Dec;18(4):313-9. doi: 10.4104/pcrj.2009.00042. PMID 19588053
- [Background] MacKenzie H, Roberts G, van Laar D, Dean T. Teenagers' experiences of living with food hypersensitivity: a qualitative study. Pediatr Allergy Immunol. 2010 Jun;21(4 Pt 1):595-602. doi: 10.1111/j.1399-3038.2009.00938.x. Epub 2009 Aug 21. PMID 19702674
- [Background] Pereira B, Venter C, Grundy J, Clayton CB, Arshad SH, Dean T. Prevalence of sensitization to food allergens, reported adverse reaction to foods, food avoidance, and food hypersensitivity among teenagers. J Allergy Clin Immunol. 2005 Oct;116(4):884-92. doi: 10.1016/j.jaci.2005.05.047. PMID 16210065
- [Background] Punekar YS, Sheikh A. Establishing the incidence and prevalence of clinician-diagnosed allergic conditions in children and adolescents using routinely collected data from general practices. Clin Exp Allergy. 2009 Aug;39(8):1209-16. doi: 10.1111/j.1365-2222.2009.03248.x. Epub 2009 Apr 17. PMID 19400899
- [Background] Tejedor-Alonso M A, Moro-Moro M, Mugica-Garcia MV. Epidemiology of Anaphylaxis: Contributions From the Last 10 Years. J Investig Allergol Clin Immunol. 2015;25(3):163-75; quiz follow 174-5. PMID 26182682
- [Background] Scadding GK, Durham SR, Mirakian R, Jones NS, Leech SC, Farooque S, Ryan D, Walker SM, Clark AT, Dixon TA, Jolles SR, Siddique N, Cullinan P, Howarth PH, Nasser SM; British Society for Allergy and Clinical Immunology. BSACI guidelines for the management of allergic and non-allergic rhinitis. Clin Exp Allergy. 2008 Jan;38(1):19-42. doi: 10.1111/j.1365-2222.2007.02888.x. PMID 18081563
- [Background] Smith HE, Wade J, Frew AJ. What proportion of adult allergy referrals to secondary care could be dealt with in primary care by a GP with special interest? Clin Transl Allergy. 2016 Jan 21;6:3. doi: 10.1186/s13601-016-0091-1. eCollection 2015. PMID 26807213
- [Derived] Hammersley V, Kelman M, Morrice L, Kendall M, Mukerjhee M, Harley S, Schwarze J, Sheikh A. Mixed-methods evaluation of a nurse-led allergy clinic model in primary care: Feasibility trial. Clin Transl Allergy. 2022 Aug;12(8):e12180. doi: 10.1002/clt2.12180. PMID 36036238